CLINICAL TRIAL: NCT04014530
Title: Study of Pembrolizumab Combined With Ataluren In Patients With Metastatic pMMR and dMMR Colorectal Adenocarcinomas or Metastatic dMMR Endometrial Carcinoma: the ATAPEMBRO Study
Brief Title: Pembrolizumab With Ataluren in Patients With Metastatic pMMR and dMMR Colorectal Carcinoma or Metastatic dMMR Endometrial Carcinoma: the ATAPEMBRO Study
Acronym: ATAPEMBRO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); PTC Therapeutics (Industry)
Responsible Party: Principal Investigator, Adriaan D. Bins, MD PhD; Principal Investigator; Oncologist, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL64152.018.18; 2017-004752-34 (EudraCT Number)
Record Dates: First submitted 2019-02-25; First posted 2019-07-10 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer; Endometrium Cancer
Keywords: Mismatch repair; Anti PD1; Immunotherapy; Metastatic disease
MeSH Terms: conditions — Colorectal Neoplasms; Endometrial Neoplasms; Neoplasm Metastasis | interventions — ataluren; pembrolizumab

STUDY DESIGN:
Intervention Model Description: In the phase-1 part of the study 2-4 groups of 3 patients each are treated with pembrolizumab 200mg i.v. q3w but with increasing ataluren doses (i.e. group1 25%, group2 50% and group3 100% of 10-10-20mg/kg). These can be either pMMR mCRC, dMMR mCRC or dMMR EC patients. The reported toxicity in phase-1 will be used to define the maximum tolerated dose (MTD) of the combination, that will determine the ataluren dose in phase-2.
  In the phase-2 part of the study a dMMR group (cohort A, 20 patients either CRC of EC) and a pMMR group (cohort B, 15 CRC patients) will be treated with pembrolizumab 200mg i.v. q3w combined with ataluren t.i.d. at the MTD defined in phase-1.
  Historic case-matched controls from the MK-3475-016 study (ClinicalTrials.gov Identifier NCT01876511) and the MK-3475-177 study (ClnicalTrials.gov Identifier NCT02563002).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Phase I dMMR and pMMR (Experimental): 2-4 groups of 3 patients treatment with 200mg i.v. Pembrolizumab q3w and dose escalation of Ataluren in order to determine the Ataluren MTD. These patients can either be pMMR/dMMR CRC and dMMR EC patients.
  Interventions: Drug: Ataluren + Pembrolizumab
- Phase II dMMR (Experimental): Mismatch repair deficient CRC or EC patients treated with 200mg i.v. pembrolizumab q3w and Ataluren at MTD.
  Interventions: Drug: Ataluren + Pembrolizumab
- Phase II pMMR (Experimental): Mismatch repair proficient CRC patients treated with 200mg i.v. pembrolizumab q3w and Ataluren at MTD.
  Interventions: Drug: Ataluren + Pembrolizumab

INTERVENTIONS:
Drug: Ataluren + Pembrolizumab — Ataluren and Pembrolizumab combination therapy

SUMMARY:
Single Center, open label, Phase I-II trial designed to test the safety and efficacy of the combination of Ataluren and Pembrolizumab for the treatment of metastatic mismatch repair deficient and proficient colorectal adenocarcinoma and metastatic mismatch repair deficient endometrial carcinoma.

DETAILED DESCRIPTION:
In controlling tumor outgrowth an intact immune surveillance is very important. PD-1 receptor-ligand interaction is a major pathway hijacked by tumors to suppress this immune control.

Pembrolizumab is a potent and highly selective humanized monoclonal antibody designed to directly block the interaction between PD-1 and its ligands and is registered for the treatment of advanced (unresectable or metastatic) melanoma of locally advanced or metastatic NSCLC in adults. In an earlier study it's effect has been shown in mismatch repair deficient tumors.

Ataluren is designed to allow the protein making apparatus (the ribosome) in cells to skip over a premature stop codon (PTC), allowing the cells to translate the sequence downstream of a premature termination codon (PTC) in mRNA transcripts. This may result in the translation of additional out-of-frame code, which is available in abundance in dMMR tumors. We argue that this may result in new target peptides for the immune-system to recognize cancer cells.

The investigators hypothesize that the formation of these peptides by Ataluren can enhance the effect of Pembrolizumab anti-PD1 therapy.

Therefore the investigators designed a Single Center, open label, Phase I-II trial designed to test the safety and efficacy of the combination of Ataluren and Pembrolizumab for the treatment of metastatic mismatch repair deficient and proficient colorectal adenocarcinoma and metastatic mismatch repair deficient endometrial carcinoma.

ELIGIBILITY:
In order to be eligible for participation in this trial, the subject must:

* Have at least one lesion with measurable disease as defined by 10mm in longest diameter for a soft tissue lesions or 15mm in short axis for a lymph node by RECIST 1.1 and irRC criteria for response assessment.
* Have received at least 1 prior cancer therapy regimen for metastatic CRC, or have refused palliative chemotherapy. In the latter case this should have been documented.
* Have a life expectancy of greater than 3 months.
* Have normal organ and marrow function as defined in protocol
* Be willing and able to provide written informed consent/assent for the trial.
* Be at least 18 years of age on day of signing informed consent.
* Be willing to provide tissue from a newly obtained pre-treatment core or excisional biopsy of a metastatic tumor lesion and the primary tumor lesion (when in place). Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible by colonoscopy or CT-guided approaches or due to safety concerns) may submit an archived specimen only upon agreement from the Sponsor.
* Be willing to provide tissue post-treatment of a core or excisional biopsy of a metastatic tumor lesion (when still in place) or of the primary tumor (when in place).
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Male subjects of childbearing potential (Section 4.7.2) must agree to use an adequate method of contraception as outlined in Section 4.7.2- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Subject must be excluded from participating in the trial if the subject:

* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 1 week prior to trial treatment.
* Has a history of prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX-40, anti-CD40, or anti-CTLA-4 antibodies.
* Has received growth factors including, but not limited to, granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), erythropoietin, etc. within 2 weeks of study drug administration. Use of such agents while on study is also prohibited. Prior use of growth factors should be documented in the patient's medical history.
* Has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has a history of any autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); CNS or motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome and Myasthenia Gravis, multiple sclerosis). Patients with thyroid disease will be allowed. Autoimmune diagnoses not listed here must be approved by the protocol chair.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or ataluren or any of their excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.
* Has received amino glucoside antibiotics within 3 days of planned start of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-Emergent Adverse Event and the determination of the maximum tolerable dose of Ataluren. | Initial dose escalation for Ataluren for first 12 pt in groups of 3, which will approximately take 1 year. All adverse events will be further reported at study compeltion: expected to be after 2 years
  To characterize toxicities and side effects of Ataluren when combined with pembrolizumab in patients with pMMR CRC, dMMR mCRC and dMMR EC. Recorded on Adverse Events form and ranking adverse event severity according to the NCI Common Terminology Criteria for Adverse Events v3.0
Objective response rate | 30 weeks
  Measured by immune-related response criteria

SECONDARY OUTCOMES:
Immune-related progression free survival | 21 weeks and 30 weeks
  irPFS
Overall survival | trough study completion: expected after 2 years.
  OS
Progression free survival | at 30 weeks
  non immune related PFS
Overall response rate | trough study completion: expected after 2 years.
  ORR
Historic case matching | trough study completion: expected after 2 years
  Historic case-matched controls from the MK-3475-016 study (ClinicalTrials.gov Identifier NCT01876511) and the MK-3475-177 study (ClnicalTrials.gov Identifier NCT02563002). Case-matching based on overall survival and immune-related response rate.

OTHER OUTCOMES:
Sequencing data comparison before and after treatment | trough study completion: expected after 4 years.
  mRNA and DNA sequencing measurements from normal blood, tumor, metastatic and polyp tissue: outcome measure will be mutations in DNA and RNA.
Identification of prediction biomarkers | trough study completion: expected after 4 years.
  Biomarker measurements from normal blood: CEA and neoantigens (peptides)
T-cell activation against neo-antigens | trough study completion: expected after 4 years.
  Elispot assays from PBMCs derived from patient blood samples to check for IFN-gamma production after peptide stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Punt, Prof., Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Adriaan D Bins, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Derived] Figaroa OJA, Spaanderman IT, Goedegebuure RSA, Cirkel GM, Jeurissen FJF, Creemers GJ, Bins AD, Tuynman J, Buffart TE. Treatment with checkpoint inhibitors for unresectable non-metastatic mismatch repair deficient intestinal cancer; a case series. BJC Rep. 2025 Sep 22;3(1):67. doi: 10.1038/s44276-025-00171-0. PMID 40983668
- See also: website sponsor — https://www.amsterdamumc.nl